CLINICAL TRIAL: NCT01621074
Title: Influence of Sodium Bicarbonate on Time-to-exhaustion at Critical Power in Endurance Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: nbc
Record Dates: First submitted 2012-06-12; First posted 2012-06-15 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Performance
MeSH Terms: interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium bicarbonate (Active Comparator)
  Interventions: Dietary Supplement: Sodium bicarbonate
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Sodium bicarbonate — Ergogenic effect
  Arms: Sodium bicarbonate
Dietary Supplement: Placebo — Placebo effect
  Arms: Placebo

SUMMARY:
During endurance exercise in the heavy and severe intensity domains, the rate at which metabolites that have been associated with the fatigue process (e.g. Pi, ADP, H, and extracellular K) accumulate increases. possibly leading to exercise cessation. Sodium bicarbonate, as a nutritional supplement, has gained attention over the past decades, because it might delay of offset fatigue. To date, there is a controversial discussion about which delivery mode (amount and frequency) might be best in optimizing endurance performance. Since the high ion load consequent to multiple ingestions might increase plasma volume, and consequently decrease bicarbonate concentrations, single acute ingestion could be more beneficial. However, in multi-day competitions or tournaments it might be necessary to use the supplement on a daily basis. Here, the investigators aim at investigating the effects of single dose or multiple dose (on five consecutive days) administration of bicarbonate vs. placebo increases endurance performance and acid-base homeostasis in trained male endurance athletes.

ELIGIBILITY:
Inclusion criteria: - male

* no cold or temperature at beginning or during the study
* between 18 and 45 years of age
* active in endurance sports (3 to 5 times per week a moderate to hart training)
* non-smoker
* no known cardiovascular or orthopedic problems
* no known limitations of kidney function
* no bearer of a cardiac pacemaker
* no medications with direct influence on the measurements. The whole intake of medicaments has to be declared in the health questionnaire by the participant.
* requirements of the health questionnaire fulfilled

Exclusion criteria: - female

* male and age under 18 or over 45 years
* cold or temperature at the beginning or during the study
* untrained (less than 3 moderate trainings per week)
* smoker
* cardiovascular or orthopedic problems
* limitations of the kidney function
* bearer of a cardiac pacemaker
* medication with direct influence on the measurements. The whole intake of medicaments has to be declared in the health questionnaire by the participant.
* requirements of the health questionnaire not fulfilled

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-10; Primary Completion 2012-08 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Time-to-exhaustion | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neurologie: Neurologische Forschung, Study Director — University Hospital Zurich, Division of Neurology; Marco Toigo, PhD, Principal Investigator — Swiss Federal Institute of Technology Zurich
Locations (1):
- University Hospital Zurich, Division of Neurology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Mueller SM, Gehrig SM, Frese S, Wagner CA, Boutellier U, Toigo M. Multiday acute sodium bicarbonate intake improves endurance capacity and reduces acidosis in men. J Int Soc Sports Nutr. 2013 Mar 26;10(1):16. doi: 10.1186/1550-2783-10-16. PMID 23531361